CLINICAL TRIAL: NCT04809272
Title: COVID-19 e-Parenting for Lifelong Health (ePLH) Pilot Study: Promoting Positive Parenting and Preventing Violence Through Online Parent Support Groups - ParentChat
Brief Title: ePLH Pilot Study: Online Support Parent Groups - ParentChat
Acronym: ePLH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Universiti Putra Malaysia (Other); Health for Youth Association, Moldova (Other); Ateneo de Manila University (Other); UNICEF Montenegro (Unknown); Alternativa (Unknown); University of Cape Town (Other)
Responsible Party: Principal Investigator, DrJamieLachman, Principal Investigator, University of Oxford
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: R72537/RE001
Record Dates: First submitted 2021-03-15; First posted 2021-03-22 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Child Maltreatment; Positive Parenting
Keywords: Parenting programme; Child physical and emotional abuse

STUDY DESIGN:
Intervention Model Description: This is a pre-post study with assessments at baseline and immediate post-intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ParentChat for parents of children ages 2-17 (Experimental): The ePLH parent support groups will be delivered over a 8 week period (i.e., 7-8 short online interactive group sessions, two per week). ePLH facilitators will moderate discussions around the parenting theme, support parents on an individual basis, and encourage them to apply the parenting skills at home. The facilitators will begin the next group engagement with a brief voice summary of the feedback and address possible solutions to 2-3 key challenges. Facilitators will also be provided with weekly supervision by an ePLH coach or trainer. A designated research assistant will provide parent support groups with needed technical support during the implementation - including IT-related support. Data bundles will be provided for internet access and to incentivise engagement.
  Interventions: Behavioral: ParentChat for parents of children ages 2-17

INTERVENTIONS:
Behavioral: ParentChat for parents of children ages 2-17 — The programme will include text/audio messages, illustrated comics, videos, and activity assignments for parents to do with their children. Parents will be prompted to give feedback regarding successes and challenges applying these parenting skills via audio or text messages during the week.

SUMMARY:
Pilot trial：

The feasibility study of the programme modules has a pre-post design with no control group, with the aims of assessing programme implementation, cultural and contextual relevance, and study feasibility. Although there will be no comparison group and it is not designed to test effects, the study also has a provisional goal of reductions in child physical and emotional abuse at immediate post-intervention.

Pre-post design:

The ePLH parent support groups will be delivered over a 8 week period (i.e., 7-8 short online interactive group sessions, two per week). The programme will include text/audio messages, illustrated comics, videos, and activity assignments for parents to do with their children. ePLH facilitators will moderate discussions around the parenting theme, support parents on an individual basis, and encourage them to apply the parenting skills at home. Parents will be prompted to give feedback regarding successes and challenges applying these parenting skills via audio or text messages during the week. The facilitators will begin the next group engagement with a brief voice summary of the feedback and address possible solutions to 2-3 key challenges. Facilitators will also be provided with weekly supervision by an ePLH coach or trainer. A designated research assistant will provide parent support groups with needed technical support during the implementation - including IT-related support. Data bundles will be provided for internet access and to incentivise engagement.

DETAILED DESCRIPTION:
Recruitment of six countries:

This study will use targeted/purposive sampling to recruit participating parents or caregivers (n = 30-100 in Malaysia, Moldova, Montenegro, North Macedonia and Philippines; 400 in South Africa). Groups will start to operate after at least 7 members have been consented and can have up to 15 members per group.

Malaysia: The National Population and Family Development Board (LPPKN) is our partner organisation for both the Semarak Kasih Parenting Program (2018-2020) and e-Semarak Kasih / ParentChat. A total of 24 staff of LPPKN have been trained for the Semarak Kasih Parenting Program, of which, 12 of them have conducted the actual program. The majority of these facilitators are University graduates holding various posts at LPPKN such as counsellors, Information Officers and Community Development Officers.

Moldova: The Health for Youth Association, has been implementing PLH for children 2-9 years in the country, in cooperation with Youth Klinics network. In Moldova, the program will be focused on caregivers/parents of adolescents (10-17 years old). The Moldovan research team will identify potential eligible parents to invite to participate in ParentChat through a) social media pages (FB, OK) of the Youth Klinics network, b) through the announcement of different partners organizations that work in social support area, and c) through the communication with YK consultants who work with parents of adolescents.

Montenegro: In Montenegro, trained facilitators from our implementing partners (health centres, kindergartens and NGOs) will recruit families by applying the same strategies used for face-to-face PLH:

* Inviting potential participants on the waiting lists for face-to-face PLH,
* Advertising on social media (the Oxford team may advertise as well if partners seek support),
* Inviting families known to service providers (e.g. parents of children attending the participating preschools, parents using psychological/mental counselling at health centres, parents users of NGO led services such as single parent support groups and the like).

North Macedonia: The Institute Alternativa - Institute for Marriage, Family and Systemic Practice has been implementing PLH for children 2-9 years in the country. The Institute Alternativa has identified potential eligible parents through the FB page of the Institute, and also those who have contacted the Institute Counselling Telephone line during the COVID-19 pandemic and expressed readiness to participate in an online programme. The psychologists who work on this help line will provide the research team with a list of eligible participants with children ages 2 to 17 years. There are already approximately 70 parents that expressed interest, of which 50 will be randomly selected for initial recruitment.

Philippines: The research team will work closely with the Department of Social Welfare and Development (DSWD) staff to identify potential eligible parents who are recipients of the conditional cash transfer program (4Ps). 4Ps staff will provide the research team with a list of eligible participants with children ages 2 to 17 years, of which 50 will be randomly selected for initial recruitment. If less than 50 of the selected participants provide consent and are eligible, the remaining adults will be randomly selected from the original list until the full target sample size is reached.

South Africa: Recruitment of programme facilitators will be done from the already trained pool of PLH facilitators in South Africa with the support of Clowns Without Borders (CWBSA). The South Africa research team and implementing team will recruit and train 10 facilitators consisting of two trained PLH trainers/Coaches from CWBSA, and 8 moderators (persons experienced in PLH implementation) who will each run 1 PSG. The two facilitators from CWBSA will also play a mentoring role for the other facilitator/moderators. The rest of the other 8 moderators will be sourced from various organisations and individuals that have been trained in PLH programmes (both PLH Kids and PLH Teens) in 5 of South Africa's provinces. For the ParentChat (Caregivers) groups, the moderators will conduct the recruitment of parents/caregivers telephonically or by one-on-one visit. This will be done from their communities where they work. Initial contact will be made with a few caregivers, who may then refer others to the group. Each group would have about 8-12 caregivers. 1000 families are expected to be reached.

ELIGIBILITY:
Inclusion criteria for participating parents or caregivers (n = 30-100 in Malaysia, Moldova, Montenegro, North Macedonia and Philippines; 500 in South Africa):

* Any person over the age of 18 years currently caring for child between the ages of 2 to 17 years
* Has regular contact with the child and spends time with the child at least two times a week
* Has access to a smartphone and is willing to join an online parenting support group to share, learn and discuss parenting
* Has provided consent to participate in the study

Inclusion criteria for facilitator and moderator (n = 10 per country):

* Age 18 or older
* Prior participation in a facilitator or moderator training workshop
* Agreement to implement the entire programme
* Provision of consent to participate in the full study

Exclusion criteria for parents or caregivers and for facilitators and moderators:

* Children below 18 years old
* Those who do not give consent to participate in the research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 522 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Child maltreatment - physical abuse and emotional abuse: ISPCAN Child Abuse Screening Tool-Intervention (ICAST-TP) - Physical and Emotional Abuse Subscales | Change between Baseline and Post (approx. 1 month after end of intervention, i.e., 3 months post pre-assessment)
  Physical abuse (including abusive discipline), emotional abuse, and neglect will be measured using 4 items from reduced version of the ISPCAN Child Abuse Screening Tool-Trial Parent version (ICAST-TP). The ICAST-TP measures parental reports of the incidence of abuse perpetrated against their child over the past month using a frequency score on a scale of 0 to 7, or 8 or more times (e.g., "In the past 4 weeks, how often did you discipline [Child Nickname] by spanking, slapping, or hitting with your hand?"). This study will assess frequency of child maltreatment for physical abuse (2 items) and emotional abuse (2 items), as well as an overall indication of previous child abuse (0 = no abuse; 1 = previous abuse).
Child maltreatment - physical abuse and emotional abuse: Frequency of overall abuse | Change between Baseline and Post (approx. 1 month after end of intervention, i.e., 3 months post pre-assessment)
  We will also assess frequency of overall abuse by summing all of the subscales as well as for each individual subscale.
Positive parenting: Parent Daily Report Checklist | Change between Baseline and Post (approx. 1 month after end of intervention, i.e., 3 months post pre-assessment)
  Two items adapted from the Parent Daily Report (PDR) will be used to assess positive parenting [19] at baseline, post-test, and every week during programme delivery. Parents will report about their behaviour within the past week instead of the past 24 hours. The two items are "how many times in the past week did you and your child do something fun together?" and "how many times in the past week did you praise your child for doing well?" The items will be rated on a frequency scale of 0 to 7, or 8 or more times.
Parenting stress: Parent Daily Report Checklist | Change between Baseline and Post (approx. 1 month after end of intervention, i.e., 3 months post pre-assessment)
  One item adapted from the Parent Daily Report (PDR) will be used to assess parenting stress [19] at baseline, post-test, and every week during programme delivery. Parents will report about their behaviour within the past week instead of the past 24 hours. The item asks, "how many times in the past week did you feel very stressed as a parent/caregiver?" The items will be rated on a frequency scale of 0 to 7, or 8 or more times.

SECONDARY OUTCOMES:
Child maltreatment - physical abuse and emotional abuse: Fortnightly Assessments | Change between T0 (baseline), T2 (2 weeks), T4 (4 weeks), T6 (6 weeks), T8 (8 weeks) and post-test at T10 (approx. 1 month after end of intervention, i.e., 3 months post pre-assessment)
  The fortnightly assessments will include a brief survey of the 7 items on primary outcomes asking parents/caregivers about how many times they engaged in positive parenting, physical and emotional abuse, and experience of parenting stress in the past 2 weeks.
Positive parenting: Fortnightly Assessments | Change between T0 (baseline), T2 (2 weeks), T4 (4 weeks), T6 (6 weeks), T8 (8 weeks) and post-test at T10 (approx. 1 month after end of intervention, i.e., 3 months post pre-assessment)
  The fortnightly assessments will include a brief survey of the 7 items on primary outcomes asking parents/caregivers about how many times they engaged in positive parenting, physical and emotional abuse, and experience of parenting stress in the past 2 weeks.
Parenting Stress: Fortnightly Assessments | Change between T0 (baseline), T2 (2 weeks), T4 (4 weeks), T6 (6 weeks), T8 (8 weeks) and post-test at T10 (approx. 1 month after end of intervention, i.e., 3 months post pre-assessment)
  The weekly assessments will include a brief survey of the 7 items on primary outcomes asking parents/caregivers about how many times they engaged in positive parenting, physical and emotional abuse, and experience of parenting stress in the past 2 weeks.
Child behaviour problems: Child and Adolescent Behaviour Inventory (CAPI) - Parent Report | Change between Baseline and Post (approx. 1 month after end of intervention, i.e., 3 months post pre-assessment)
  Child behaviour problems will be measured using the Child and Adolescent Behaviour Inventory (CABI). The CABI assesses a wide range of internalizing and externalizing symptoms in children and adolescents and is relatively shorter than the Child Behaviour Check List (CBCL), making it a practical and reliable tool for measuring behaviour problems. Parents report on their child's behaviour during the past week. The irritability subscale and the externalizing subscale will be used to measure problem behaviours. Items on both subscales are summed to create a total score of child behaviour problems.
Child behaviour problems: Three Problem Rating Scale - Parent Report | Change between Baseline and Post (approx. 1 month after end of intervention, i.e., 3 months post pre-assessment)
  2 items adapted from the Three Problem Scale-Parent Report will be used to assess whether specific concerns or issues parents are having with their children change during an intervention. Parents report whether the behaviour has occurred in the past week and select the most problematic behaviour from the list of 10 and indicate how challenging the behaviour was on a scale of 0 to 8 (0 = not a problem, 8 = could not be worse).
Sexual abuse risk: Parent Report | Change between Baseline and Post (approx. 1 month after end of intervention, i.e., 3 months post pre-assessment)
  One item will be used to assess parents' perceptions of reduction of sexual abuse risk. The item asks, "how confident do you feel you are to protect your child from sexual abuse online or in-person?" Parents/primary caregivers will respond based on an 8-point Likert scale of 0 to 4 (0 = Not confident at all; 8 = Extremely confident).
Attitude toward punishment: Multiple Indicator Cluster Survey (MICS) 5 Child Discipline module - Parent Report | Change between Baseline and Post (approx. 1 month after end of intervention, i.e., 3 months post pre-assessment)
  Attitudes toward punishment will be assessed using one item from the UNICEF Multiple Indicator Cluster Survey (MICS) 5 Child Discipline module. The MICS item asks the parent/primary caregiver: "In order to bring up, raise up, or educate a child properly, the child needs to be physically punished." Parents/primary caregivers will report whether they disagree or agree with the statement.
Parent well-being: Depression, Anxiety, and Stress Scale (DASS) - Parent Report | Change between Baseline and Post (approx. 1 month after end of intervention, i.e., 3 months post pre-assessment)
  The depression subscale of the Depression, Anxiety, and Stress Scale (DASS) will assess caregiver well-being. The DASS is a 21-item scale used as a screening tool to measure depression, anxiety, and stress in adults. The stress subscale includes 7 items (e.g., ""I felt down-hearted and sad"). Caregivers report on the frequency of depressive symptoms in the previous week using a Likert scale (0 = Never, 1 = Sometimes, 2 = Often, 3 = Always).
Parent exposure to IPV and intimate partner coercion: WHO Multi-Country Questionnaire on Women's Health and Domestic Violence against Women (WHO) - Parent Report | Change between Baseline and Post (approx. 1 month after end of intervention, i.e., 3 months post pre-assessment)
  Adult self-report of experiencing intimate partner violence and coercion over the past week will be assessed using 2 items from an adapted version of the Revised Conflict Tactics Scale Short Form (CTS2S). The CTS2S scale includes 2 items on the frequency of physical assault ("partner pushed, shoved, or slapped me"), and psychological aggression ("partner insulted, shouted, yelled, or swore at me"). All answers are coded on a frequency scale of 0 to 7, or 8 or more times. Alternatively, caregivers will indicate whether they experienced violence from a partner (e.g., hitting, pushing or slapping; insulting, shouting or yelling) in the past week by answering yes or no.
Parent exposure to IPV and intimate partner coercion: Revised Conflict Tactics Scale Short Form (CTS2S) | Change between Baseline and Post (approx. 1 month after end of intervention, i.e., 3 months post pre-assessment)
  Adult self-report of experiencing intimate partner violence and coercion over the past week will be assessed using 2 items from adapted items from the WHO Multi-Country Study Questionnaire on Women's Health and Life and Domestic Violence against Women (WHO). The adapted WHO questionnaire includes 2 items on coercion and emotional violence ("my partner insisted on knowing where I was at all times"), and on restriction of financial autonomy (e.g., "my partner refused to give me money for household expenses, even when he/she had money for other things."). All answers are coded on a frequency scale of 0 to 7, or 8 or more times. Alternatively, caregivers will indicate whether they experienced violence from a partner (e.g., hitting, pushing or slapping; insulting, shouting or yelling) in the past week by answering yes or no.

OTHER OUTCOMES:
Sociodemographic information: UNICEF Multiple Indicators Cluster Survey (MICS) Household Survey | Baseline
  Basic caregiver and child demographic information will be asked using items from the UNICEF Multiple Indicators Cluster Survey (MICS) Household Survey. The MICS was developed to monitor the situation of children and women on a global level and is based on Demographic and Health Surveys. It has been used widely throughout low- and middle-income countries (LMIC) including the Philippines. It assesses caregiver/child age, gender, marital status, education level, basic literacy, child's relationship to caregiver, and the presence of other caregivers in the household. It also assesses other household socio-demographic characteristics including whether or not the family receives any government grants. Demographic questions will be included in the baseline assessments. Items on marital status, household size, presence of other caregivers in the household, government assistance, and education level will be included in the intake survey administered by facilitators or moderators after baseline
COVID-19 information: Parent Report | Baseline
  One item will ask parents to indicate how COVID-19 affected their family using 6 options (someone in my family has had COVID-19 symptoms, someone in my family has died of COVID-19, my family has been experiencing financial stress due to COVID-19, family has been experiencing emotional stress due to COVID-19, my family has not been negatively affected by COVID-19, my family has not been affected by COVID-19). This item will be administered by facilitators or moderators in the intake survey after baseline assessment.
Implementation Fidelity: Facilitator check-lists | Post (approx. 1 month after end of intervention, i.e., 3 months post pre-assessment)
  Implementation fidelity of the ePLH programme will be measured using self-report checklists by facilitators to examine the extent to which core intervention components are delivered. These checklists will include specific activities for each session, such as home practice discussion and role-playing exercises. Then, in order to produce a basic level of fidelity, a ratio of programme implementation to programme design will be created for the self-report scores. According to Borrelli and colleagues, a standard of 80% programme fidelity will be considered as "high treatment fidelity".
Programme Adherence - Enrolment rates: Attendance registration | Post (approx. 1 month after end of intervention, i.e., 3 months post pre-assessment)
  Programme adherence will be assessed by examining rates of enrolment, attendance, and dropout. Enrolment rates will be based on the number of parents who participated in the programme. Parents are considered to have participated in the programme if they sent at least one message on the online PSG platform.
Programme Adherence - Mean attendance rates: Attendance registration | Post (approx. 1 month after end of intervention, i.e., 3 months post pre-assessment)
  Programme adherence will be assessed by examining rates of enrolment, attendance, and dropout. Mean attendance rates for enrolled participants will be determined based on the ratio of number of attended sessions to the total number of programme sessions.
Programme Adherence - Dropout rates: Attendance registration | Post (approx. 1 month after end of intervention, i.e., 3 months post pre-assessment)
  Programme adherence will be assessed by examining rates of enrolment, attendance, and dropout. Dropout rates for enrolled participants will be defined as the percentage of participants who fail to attend at least two consecutive sessions and do not attend any sessions at a later stage.
Participant satisfaction: Parent overall satisfaction | Post (approx. 1 month after end of intervention, i.e., 3 months post pre-assessment)
  Participant satisfaction will be examined for parents/caregivers who attend at least one session of the programme. At post-intervention, participants will report on 4 items drawn from a Parent Satisfaction Survey asking about their satisfaction with the programme. Mean and standard deviation scores will be calculated for the overall participation satisfaction scale (1 = Very unhelpful; 5 = Very helpful).
Facilitator and participant engagement: Process monitor reports | Once per week over 8 week during programme delivery
  Engagement will be based on the number of messages, type of messages (text/audio/video), and length of messages (word count) sent to the online PSGs by facilitators and participants for each session. It will also be indicated by the number of activities completed by each participant (e.g., home assignments). Process monitors present in online PSGs will export message logs and accomplish a weekly report that includes a summary of issues or challenges that were observed regarding facilitators' and participants' engagement. Content or narrative analysis of text messages will be conducted to further investigate acceptability of programme content, quality of programme delivery, and patterns of communication and interaction between facilitators, moderators and participants.
Acceptability - Participants' observed change in parent-child relationships at home during programme: Focus groups | Post (approx. 1 month after end of intervention, i.e., 3 months post pre-assessment)
  Participants' observed change in parent-child relationships at home during programme will be assessed by conducting focus groups with facilitators and moderators (n = 10). FGDs with facilitators and moderators will last approximately 60 minutes and will be conducted via a video conference platform (e.g., Microsoft Teams).
  Online focus groups will be recorded with written notes as a backup. All data will be transcribed verbatim and will be translated into English and back-translated into local languages to verify accuracy. Qualitative data obtained from focus groups will be analysed using a thematic analysis approach with open, axial, and selective coding.
Acceptability - Cultural acceptability and appropriateness of programme materials, delivery, and key programme components: Focus groups | Post (approx. 1 month after end of intervention, i.e., 3 months post pre-assessment)
  Cultural acceptability and appropriateness of programme materials, delivery, and key programme components will be assessed by conducting focus groups with facilitators and moderators (n = 10). FGDs with facilitators and moderators will last approximately 60 minutes and will be conducted via a video conference platform (e.g., Microsoft Teams).
  Online focus groups will be recorded with written notes as a backup. All data will be transcribed verbatim and will be translated into English and back-translated into local languages to verify accuracy. Qualitative data obtained from focus groups will be analysed using a thematic analysis approach with open, axial, and selective coding.
Acceptability - Existing barriers to participation during sessions and engagement in home practice and other activities: Interviews | Post (approx. 1 month after end of intervention, i.e., 3 months post pre-assessment)
  Existing barriers to participation during sessions and engagement in home practice and other activities will be assessed by conducting interviews with programme participants (n = 10-12). Participants will be purposively selected with the inclusion criteria of attending at least one session. Selection will be based on those with high engagement (n = 3-4), those with low engagement (n = 3-4), those who dropout (n = 3-4).
  Trained researchers will conduct all of the interviews with parents in local languages. Interviews with participants will last approximately 30 minutes and will be conducted over the phone.
  Phone interviews will be recorded with written notes as a backup. All data will be transcribed verbatim and will be translated into English and back-translated into local languages to verify accuracy. Qualitative data obtained from interviews will be analysed using a thematic analysis approach with open, axial, and selective coding.
Feasibility of Programme for scale-up: Weekly facilitator survey - Facilitator Report | Once per week over 8 week during programme delivery
  Quantitative data concerning the feasibility of ePLH for scale-up will be assessed through a weekly facilitator survey, which will indicate how much time they spend on chat sessions (e.g. "please enter the time that the chat session began on Day 1" and "please enter the time the chat session ended on Day 1") and coaching sessions (e.g. "how long in minutes did you spend preparing for the second chat session on Day 5?") and briefly describe the interaction between them and participants.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie M. Lachman, DPhil, Principal Investigator — University of Oxford; Rumaya Juhari, PhD, Principal Investigator — University Putra Malaysia; Galina Lesco, PhD, Principal Investigator — Health for Youth Association, Moldova; Ida Ferdinandi, PhD, Principal Investigator — UNICEF Montenegro; Marija Raleva, PhD, Principal Investigator — Alternativa; Rosanne Jocson, PhD, Principal Investigator — Ateneo de Manila University; Kufre Okop, PhD, Principal Investigator — University of Cape Town
Locations (1):
- University of Oxford, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data will be shared on Open Science Framework after the completion of the study and results are published
Supporting Information: Study Protocol
Time Frame: Indefinitely
Access Criteria: Accessibility of the data will require approval from the study team. The study investigators, led by the PI, will jointly make decisions on whether to supply research data to potential new users. Research data will be deposited in and available in the UK Data Archive solely for non-profit use.